CLINICAL TRIAL: NCT03770078
Title: Assessment of New Enhanced Ostomy Device in Real-life Settings in Subjects Having a Stoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP300
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Ileostomy - Stoma; Colostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study period (Experimental): First the subjects will use the comparator (SenSura Mio) and then the test products (Test Product A)
  Interventions: Device: Test Product A

INTERVENTIONS:
Device: Test Product A — The test product is a newly developed ostomy product

SUMMARY:
The study investigates the performance of a new adhesive with regard to the skin condition

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have an ileostomy or a colostomy with liquid* output (as their usual output)
* Be at least 18 years of age and have full legal capacity
* Have had their stoma for at least three months
* Be able to use products with max cut size 45 mm
* Have self-reported problems with leakage** (three times within 14 days)
* Handle the Clinical App, test product and comparator product themselves
* Use a flat SenSura® Mio or a flat SenSura® with standard adhesive as their current product
* Minimum change of baseplate at least once every 3rd day
* Are willing and suitable (determined by investigator/study nurse) to use the test product and comparator without using a paste/mouldable ring during the investigation
* Are willing and suitable (determined by investigator/study nurse) to use a 1-piece product during the investigation

Exclusion Criteria:

* Are currently receiving or have within the past two months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis)
* Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area (e.g. lotion or spray) or systemic treatment* (e.g. injection or tablets).
* Get a positive result of a pregnancy test for women of childbearing age/fertile (**clarified in section 6.3.2)
* Are breast feeding
* Are participating in other interventional clinical investigations or have previously participated in this investigation

Exception:

Participation in other Coloplast in-house clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP300) protocol.

- Have known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Consultant
Locations (4):
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - Coloplast, Humlebæk
  - CCBR Vejle, Vejle
- KTA Prim Stockholm, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline and Test Period: The users tested a product for two weeks (baseline) and then went on to try the Test Product A for 28 days.
Period: Overall Study
Arm/Group | Baseline and Test Period
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Baseline and Test Period
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 23
Region of Enrollment [Number; unit: participants]
  Sweden | 4
  Denmark | 19

OUTCOME MEASURES:

1. Primary Outcome: Trans Epidermal Water Loss
Description: Trans epidermal water loss is an objective skin measurement that is measures the evaporation of water on the skin surface using a probe (DermaLab).The trans epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin due to evaporation. When the skin barrier is damaged this evaporation of water increases. Thus, transepidermal water loss can be used to assess skin damage.
  Trans Epidermal Water Loss is reported in grams of water per square meter per hour (g/m^2/h).
Time Frame: Four weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: g/m^2/h
Groups:
- Comparator Product: The users tested a product for two weeks (baseline)
- Test Product A: Tested test product A for 28 days
Arm/Group | Comparator Product | Test Product A
Number analyzed (Participants) | 23 | 23
g/m^2/h | 39.0 [32.6 to 46.6] | 35.9 [30.1 to 42.7]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Groups:
- Baseline/Comparator Product: The users tested a product for two weeks (baseline)
- Test Product A: Test Product A was used for 28 days.
Arm/Group | Baseline/Comparator Product | Test Product A
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/23 | 5/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline/Comparator Product (N=23) | Test Product A (N=23)
Peristomal skin complications (Skin and subcutaneous tissue disorders) | 3 (5) | 4 (7)
Swollen stoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased stoma mucous production (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03770078/Prot_SAP_000.pdf